CLINICAL TRIAL: NCT07139587
Title: The Efficacy and Safety of Iparomlimab/Tuvonralimab (Anti PD-1/CTLA-4) Combined With Albumin-bound Paclitaxel in Second-line Treatment of Patients With Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qingxia Li (Other)
Responsible Party: Sponsor-Investigator, Qingxia Li, Professor, Hebei General Hospital
Organization: Hebei General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-399
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Immunotherapy; gastric cancer; gastroesophageal junction adenocarcinoma; PD-1/CTLA-4
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab combined with albumin-paclitaxel (Experimental): Iparomlimab and Tuvonralimab: 5.0mg/kg, D1, Q3w; Albumin-paclitaxel: 260mg/m², D1, Q3w
  Interventions: Drug: Iparomlimab/Tuvonralimab (anti PD-1/CTLA-4) combined with albumin-bound paclitaxel

INTERVENTIONS:
Drug: Iparomlimab/Tuvonralimab (anti PD-1/CTLA-4) combined with albumin-bound paclitaxel — Iparomlimab/Tuvonralimab : 5.0mg/kg, D1, Q3W Albumin-bound paclitaxel: 260mg/m², D1, Q3W

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab (anti PD-1/CTLA-4) combined with albumin-paclitaxel in the second-line treatment of patients with advanced gastric/gastroesophageal junction adenocarcinoma. The main questions it aims to answer are: 1. Can the combination of Iparomlimab/Tuvonralimab and albumin-paclitaxel for advanced gastric cancer/gastroesophageal junction cancer who has progressed or is intolerant to first-line SOC prolong the PFS and OS, improve ORR, DCR, and prolong DoR; 2. Whether Iparomlimab/Tuvonralimab ( anti PD-1/CTLA-4) combined with albumin-paclitaxel for second-line treatment remains effective for patients who have progressed from first-line PD-1±chemotherapy; 3. The safety and tolerability of Iparomlimab/Tuvonralimab in combination with albumin-paclitaxel for second-line treatment.Participants will:1. Use Iparomlimab/Tuvonralimab 5.0mg/kg, D1, Q3W; At least 30 minutes later, administer the chemotherapy albumin-paclitaxel: 260mg/m², D1, Q3W, and complete the infusion within 30 minutes. The combined regimen was administered every 3 weeks, with efficacy evaluated every 2 cycles (RECIST 1.1) until disease progression, intolerable toxicity or patient withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75;
* ECOG PS 0-2;
* Histologically confirmed advanced of the gastric cancer/gastroesophageal junction adenocarcinoma;
* Failure of first-line treatment: Progression or intolerance after receiving platinum-based (oxaliplatin/cisplatin) + fluorouracil (5-FU/ capecitabine /S-1) regimens;
* The first-line use of PD-1 inhibitors is permitted;
* At least one measurable lesion (RECIST v1.1);
* Good organ function (ANC≥1.5×109/L, PLT≥100×109/L, with normal liver and kidney functions）.

Exclusion Criteria:

* Her2-positive gastric cancer/gastroesophageal junction adenocarcinoma;
* Active autoimmune disease;
* Previously received PD-1/CTLA-4 bispecific antibody or taxanes at first-line treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | 3 years
  Assessed by INV based on RECIST 1.1, defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall survival（OS） | 4 years
  Defined as the time between the date of enrollment and the date of death (by any cause).
Objective response rate（ORR） | 3 years
  Defined as the percentage of participants whose BOR is either a confirmed CR or PR（assessed by INV based on RECIST 1.1）
Disease control rate（DCR） | 3 years
  Defined as the percentage of participants who have a BOR of CR, PR, SD, or NON-CR/NON-PD（assessed by INV based on RECIST 1.1）
Duration of Responce （DoR） | 4 years
  Defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression or death due to any cause, whichever occurs first（assessed by INV based on RECIST 1.1）
Adverse events | 4 years
  Incidence of AEs, SAEs, deaths and laboratory abnormalities in all treated participants

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei General Hospital, Shijiazhuang, Hebei, China